CLINICAL TRIAL: NCT04684030
Title: The Management of Glucose Control and Hypoglycemic Prevention Using Continuous Glucose Monitoring System in Patients With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0831
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring; Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled, single-center clinical study. Patients will randomized 1:1 to either CGMS or conventional self-monitoring of blood glucose (SMBG) group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGMS group (Experimental): Using continuous glucose monitoring system(CGMS) group
  Interventions: Device: Continuous glucose monitoring system(CGMS)
- SMBG group (Active Comparator): Self-monitoring of blood glucose group (conventional fingerpricking method)
  Interventions: Device: Self-monitoring of blood glucose (conventional fingerpricking method)

INTERVENTIONS:
Device: Continuous glucose monitoring system(CGMS) — Patients will randomized 1:1 to either continuous glucose monitoring system(CGMS) or conventional self-monitoring of blood glucose (SMBG) group. After the randomization, patients in CGMS group will given education on how to use the device and check the result using the smart phone. The data collected from the sensors were computed to generate the respective ambulatory glucose profiles so as to determine the total numbers of scans conducted during the study period.
  Arms: CGMS group
Device: Self-monitoring of blood glucose (conventional fingerpricking method) — Patients will randomized 1:1 to either continuous glucose monitoring system(CGMS) or conventional self-monitoring of blood glucose (SMBG) group. After the randomization, patients in SMBG group will check their blood glucose by finger pricking method and record the data in a notebook to share the data in their outpatient clinic visit.
  Arms: SMBG group

SUMMARY:
This study was designed to evaluate the glucose control and hypoglycemic prevention effect of using continuous glucose monitoring system(CGMS) in patients with type 1 diabetes. This is a prospective randomized controlled, single-center clinical study. Patients will randomized 1:1 to either CGMS or conventional self-monitoring of blood glucose (SMBG) group. After 12 weeks of applying the CGMS sensors, the improvement of parameters collected from the CGMS will be estimated in comparison with data collected from the SMBG.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ages >= 20 years
2. Patients diagnosed with type 1 diabetes.
3. Patients with glycated hemoglobin (HbA1c) > 8.0% within 6 months before screening
4. Patients who agree to perform self blood glucose monitoring responsibly during the study period
5. Patients diagnosed with type 1 diabetes minimum 3 months prior to recruitment

Exclusion Criteria:

1. Patients diagnosed with type 2 diabetes.
2. Patients with chronic disease (Excluding thyroid disorders in which thyroid function is controlled in the normal range), or psychiatric disease
3. Patients who cannot use the device properly such as an illiterate person or foreigners
4. Patients incapable of making decisions based on their own judgement and will
5. A person who may not participate in the study according to investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
The change of glycated hemoglobin (HbA1c) level | 12 weeks after applying continuous glucose monitoring system
  The HbA1c levels in this study will analyzed twice during the study, once at the baseline and after the CGMS testing was initiated. The improvement of HbA1c level in CGMS group will be estimated and compare it with the change in HbA1c level in the SMBG group.

SECONDARY OUTCOMES:
The number of participants with improved clinical glycometabolic parameters | 12 weeks after applying continuous glucose monitoring system
  Clinical glycometabolic parameters (HbA1c, glycated albumin, glycemic variability, hypoglycemia, calculated insulin dose, patient's self confidence in diabetes self-care, Quality of life) and anthropometric parameters (Blood pressure, Body weight, BMI etc)

CONTACTS AND LOCATIONS:
Overall Officials: EunSeok Kang, Ph.D, Principal Investigator — Severance Hospital Diabetes Center
Locations (1):
- Severance Hospital Diabetes Center, Division of Endocrinology and Metabolism, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No